CLINICAL TRIAL: NCT06196138
Title: The Effect of Chewing Gum and Hot Compresses on Postoperative Pain, Bowel Function, and Patient Comfort After Gynecologic Oncologic Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Chewing Gum and Hot Compresses on Gynecologic Oncologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University (Other); Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Eda Polat, Research Asisstant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulMU20
Record Dates: First submitted 2023-12-22; First posted 2024-01-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-03

CONDITIONS: Gynecologic Nursing; Pain
MeSH Terms: conditions — Pain | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gum (Experimental): Patients who will chew gum after surgery will constitute this group
  Interventions: Other: Gum
- Hot Compress (Experimental): Patients who will undergo hot compress after surgery will constitute this group
  Interventions: Other: Hot Compress
- Control (No Intervention): Patients who will undergo routine protocol will constitute this group

INTERVENTIONS:
Other: Gum — In the postoperative period, starting from the 4th hour, chewing gum is done 3 times a day, morning, noon and evening, for 30 minutes each, until the patient passes the first flatus.
  Arms: Gum
Other: Hot Compress — Starting from the 1st postoperative day, patients will receive hot application (to the lumbar region) for 10 minutes in the morning and evening. The hot application is applied by wrapping 2 towels in a water bag containing 55 ± 2 °C hot water. The water bag is applied to the lumbar region for 10 minutes with the patient in the supine position. The application is continued until the patient passes the first flatus.
  Arms: Hot Compress

SUMMARY:
The passage discusses the recovery of gastrointestinal (GI) function after abdominal surgery and the potential impact on patient comfort. After surgery, small bowel activity typically returns to normal within a few hours, gastric activity within 24-48 hours, and colonic activity within 48-72 hours. However, the delayed mobility of the GI system postoperatively can lead to issues such as abdominal bloating, nausea, vomiting, and pain. These symptoms can negatively affect patient comfort, leading to increased post-operative pain, decreased mobility, reduced satisfaction, and a longer hospital stay. Therefore, interventions that expedite the normalization of bowel activity are crucial. Chewing is suggested to stimulate intestinal motility by activating the cephalovagal pathway, which influences neurogenic and hormonal factors regulating GI functions. Postoperative heat application aims to prevent hypothermia, enhance bodily functions, and potentially promote bowel motility by stimulating somatic nerves. The study explores the effects of gum chewing and hot application protocols on postoperative pain, bowel function, and patient comfort after gynecologic oncologic surgery. It aims to contribute valuable insights to the existing literature on postoperative outcomes.

DETAILED DESCRIPTION:
After abdominal surgery, small bowel activity returns to normal within a few hours, gastric activity within 24-48 hours, and colonic activity within 48-72 hours. Due to the delayed mobility of the gastrointestinal (GI) system in the postoperative period, gas and secretions accumulated in the stomach and intestines cause abdominal bloating, nausea, vomiting, and pain, negatively impacting patient comfort. This can lead to increased post-operative pain, decreased post-operative mobility, decreased patient satisfaction and prolonged hospital stay. Therefore, procedures that shorten the time to normalization of bowel activity in the postoperative period are very important. Chewing stimulates intestinal motility in humans. The chewing mechanism is thought to work by stimulating the cephalovagal pathway. Stimulation of the cephalovagal pathway stimulates various neurogenic and hormonal factors that modulate the functions of the gastrointestinal tract. Problems related to decreased intestinal motility after minimally invasive surgery can cause postoperative side effects due to delayed recovery of GI function. The basic rationale of postoperative heat application is to prevent the development of hypothermia during and after surgery by regionally warming the patient's body, eliminating the slowing effect of hypothermia, and helping to activate bodily functions early. It has been suggested that heat application may reflexively promote bowel motility by stimulating somatic nerves via the supraspinal or spinal cord, and it has been demonstrated that stimulation of warm receptors in the skin with heat may reflexly inhibit sympathetic nerves and promote parasympathetic nerve activity in the bowel as a supraspinal and spinal reflex. There are few studies in the literature examining the effect of chewing gum and heat application on postoperative outcomes after gynecologic oncologic surgery. No study was found that compared the two applications. This study was designed to compare the effects of gum chewing and hot application protocols on postoperative pain, bowel function, and patient comfort after gynecologic oncologic surgery. It is believed that this study will make an important contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* To undergo elective minimally invasive gynecologic surgery
* No cognitive, affective and mental problems that would prevent gum chewing and hot application
* Does not have any chronic disease
* No previous abdominal surgery
* Turkish speaking and
* Women who volunteer to participate in the study will be included.

Exclusion Criteria:

* Who wants to leave the work for any reason
* History of ileostomy and colostomy
* He was taken to intensive care after the surgery and
* Women with postoperative complications (bleeding, infection, etc.) will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients of the female gender will be included, as they are patients undergoing gynecological surgery.
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 8 months
  This scale, which can be used horizontally or vertically, is shaped like a 10 cm line. The scale begins with "No pain" and ends with "My pain is very severe. The person is asked to select a number between 0 and 10 that corresponds to the pain they feel on this scale.
General Comfort Scale | 8 months
  The highest total score that can be obtained from the scale is 192 and the lowest total score is 48. Obtained The total score depends on the number of scale items.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Beke, MSc, Principal Investigator — Dr. Abdurrahman Yalcin Training and Research Hospital
Locations (1):
- Dr. Abdurrahman Yalcin Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision will be made by the researchers at the end of the research.

REFERENCES:
- [Background] Akladios C, Darai E, Golfier F, Lecuru F, Collinet P, Uzan C, Lavoue V, Guyon F, Ferron G, Querleu D. [National certification for gynecological cancer surgery]. Bull Cancer. 2021 Sep;108(9):806-812. doi: 10.1016/j.bulcan.2021.03.019. Epub 2021 Jun 30. French. PMID 34217437
- [Background] Schneider S, Armbrust R, Spies C, du Bois A, Sehouli J. Prehabilitation programs and ERAS protocols in gynecological oncology: a comprehensive review. Arch Gynecol Obstet. 2020 Feb;301(2):315-326. doi: 10.1007/s00404-019-05321-7. Epub 2019 Oct 15. PMID 31616986
- [Background] Nanthiphatthanachai A, Insin P. Effect of Chewing Gum on Gastrointestinal Function Recovery After Surgery of Gynecological Cancer Patients at Rajavithi Hospital: A Randomized Controlled Trial. Asian Pac J Cancer Prev. 2020 Mar 1;21(3):761-770. doi: 10.31557/APJCP.2020.21.3.761. PMID 32212805
- [Background] Yin YN, Xie H, Ren JH, Jiang NJ, Dai L. The impact of gum-chewing on postoperative ileus following gynecological cancer surgery: A systematic review and meta-analysis of randomized controlled trials. Front Oncol. 2023 Jan 17;12:1059924. doi: 10.3389/fonc.2022.1059924. eCollection 2022. PMID 36733360
- [Background] Phutsisen J, Kietpeerakool C, Jampathong N, Chumworathayi B, Temtanakitpaisan A, Aue-Aungkul A, Boontasaeng P. Effects of Cassia alata Linn on bowel function recovery following surgery for gynecological cancer: A randomized controlled trial. Complement Ther Med. 2019 Dec;47:102222. doi: 10.1016/j.ctim.2019.102222. Epub 2019 Oct 21. PMID 31779993